CLINICAL TRIAL: NCT05429190
Title: Validation of a Short and Effective MRI Surveillance (SMS) Protocol for Hepatocellular Carcinoma Screening in Practice
Brief Title: Validation of SMS Protocol for HCC Screening in High-risk Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Céline van de Braak, PhD-student, Erasmus Medical Center
Other Study IDs: 2021-2 / 13803
Record Dates: First submitted 2022-06-14; First posted 2022-06-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Cirrhosis; Hepatitis; Hepatocellular carcinoma; MRI; Surveillance
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis; Hepatitis | interventions — Spermine Synthase; Clinical Protocols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Short MRI surveillance (SMS) protocol — Bi-annual, non-contrast agents, MRI screening consisting of Diffusion Weighted Imaging (b-values of 50 and 800 s/mm2), T2-weighted imaging and T1-weighted in- and out-of-phase imaging
Radiation: Bi-annual ultrasonography screening — Bi-annual ultrasonography for screening of HCC in high-risk patients

SUMMARY:
The investigators will assess implementation of the proposed SMS protocol as a surveillance tool in patients at high risk of developing HCC in a prospective multicenter study.

DETAILED DESCRIPTION:
Over the past 20 years, the prevalence of HCC has been growing extensively. HCC makes up for 75-85% of primary liver cancers and has a poor prognosis with a 5-year survival rate lower than 20%. The incidence of HCC is higher in patients diagnosed with hepatitis and/or cirrhosis. The current guidelines recommend a bi-annual US screening of this patient group. However, recent meta-analysis showed that the sensitivity of such US surveillance for detecting early stage HCC is merely 47%. In addition, early detection of small HCC lesions (with a diameter less than 2 cm) will provide a higher survival chance. It is therefore of major importance to develop a better surveillance tool.

The use of MRI should be considered as a surveillance tool for this patient group. In comparison to US, MRI come with high cost, long duration of the scan, limited availability and a potential risk related to the use of contrast agents. The investigators have developed and validated a short MRI surveillance (SMS) protocol for HCC screening in high-risk patients. This protocol has been evaluated among a database of 215 patients. In this prospective, multicenter study, the investigators will evaluate the value of the SMS protocol in a high-risk patient group and they will assess the cost-effectiveness of the SMS protocol as a surveillance tool with respect to a bi-annual US screening.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients above 18 years of age
* High-risk patients with cirrhosis and/or hepatitis

Exclusion Criteria:

* Patients below the age of 18 years
* Patients who will not sign the informed consent form
* Patients with general contra-indications for undergoing MRI examination

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with high-risk (cirrhosis and/or hepatitis) of developing HCC conform Dutch guidelines for HCC surveillance (https://www.oncoline.nl/hepatocellulair-carcinoom)
Sampling Method: Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Increased sensitivity for HCC detection | 3 years
  Detection of HCC using the SMS protocol will be compared to US surveillance

SECONDARY OUTCOMES:
Cost-effectiveness analysis of SMS protocol | 2 years
  A cost-effectiveness analysis will be performed for the SMS protocol by measuring all direct medical costs. Using a Markov Model, the final outcome will give us an incremental cost-effectiveness ratio. Although direct costs of MRI (SMS protocol) are higher than US, improved detection of early HCC with SMS may finally prove more cost-effective than US

OTHER OUTCOMES:
Patients acceptance of the SMS protocol (through a questionnaire) | 3 years
  Patients will be invited to circumvent their personal experiences, including confidence with both the SMS and US. The outcome may prove patients acceptance of SMS as the new standard for HCC surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. de Man, Principal Investigator — Erasmus Medical Center; Dr. Takkenberg, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Prof. Dr. Uyl-de Groot, Principal Investigator — Erasmus School of Health Policy & Management Rotterdam; Prof. Dr. IJzermans, Principal Investigator — Erasmus Medical Center; Dr. Bos, Principal Investigator — Erasmus Medical Center
Locations (6):
- Netherlands (6):
  - Academic Medical Center, Amsterdam, North Holland
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - St. Franciscus Gasthuis & Vlietland, Rotterdam, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland